CLINICAL TRIAL: NCT01739387
Title: A Randomised, Open-label, Cross-over Study of Flutiform® BAI and Flutiform® pMDI Devices in Adolescents and Adult Subjects With Persistent Asthma or Chronic Obstructive Pulmonary Disease (COPD) to Assess Patient Handling.
Brief Title: A Study Assessing Patient Handling of Flutiform® Breath-Actuated Inhaler (BAI) and Flutiform® Pressurised Metered Dose Inhaler (pMDI)
Status: Completed | Type: Observational
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: KFL9501
Record Dates: First submitted 2012-11-14; First posted 2012-12-03 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Asthma; COPD
Keywords: Flutiform®; Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breath actuated inhaler (BAI): Placebo. Two to nine puffs on one day only
  Interventions: Device: Flutiform® pMDI and Breath Actuated Inhaler (BAI)
- Flutiform® pMDI: Placebo. Two to nine puffs on one day only
  Interventions: Device: Flutiform® pMDI and Breath Actuated Inhaler (BAI)

INTERVENTIONS:
Device: Flutiform® pMDI and Breath Actuated Inhaler (BAI) — Both devices contain placebo

SUMMARY:
This study will compare the patient handling of Flutiform® pMDI (pressurised metered dose inhaler) and a breath activated device (BAI). Patient handling will be assessed using assessment criteria which detail the correct handling steps for each inhaler.

DETAILED DESCRIPTION:
Approximately 340 subjects aged 12 years and over who have asthma or chronic obstructive pulmonary disease (COPD), and are on medication for their condition will be recruited for the study. Subjects will be recruited to ensure that different severities of disease are included in the study.

Severity of disease will be determined by predicted FEV1. During the study subjects will be trained to use both the pMDI device and the BAI device being compared. Following training the subjects' use of each device will be assessed by a trainer/assessor using assessment criteria which cover handling, actuation and inhalation aspects for each of the devices under test. The order in which subjects receive each device will be determined using a randomisation schedule.

During the study subjects will continue to take their prescribed asthma or COPD medication. The pMDI and BAI devices used for the patient handling assessment will only contain placebo.

The duration of the study for a subject will be up to 58 days. Training and use of each device will be separated by 7 to 21 days

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent.
2. Male and female subjects ≥12 years old.
3. Documented history of asthma or COPD for ≥ 6 months prior to screening visit.
4. Subjects receiving ICS and LABA
5. Can perform spirometry adequately.
6. Willing and able to attend all study visits

Exclusion Criteria:

1. Any severe chronic respiratory disease other than asthma and COPD.
2. Evidence of a clinically unstable disease as determined by medical history or physical examination that, in the Investigator's opinion, precludes entry into the study or may confound between-period comparisons. 'Clinically unstable' is defined as any disease that, in the opinion of the Investigator, would put the Subject at risk through study participation.
3. Any serious neuromuscular disorder, or orofacial disease preventing the application of an inhaler to the mouth.
4. Known sensitivity to inhaler propellant or excipients.
5. Participation in a clinical drug study within 30 days of the screening visit.
6. Current participation in a clinical study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthmas and COPD patients aged 12 and above obtained from primary care and advertising in Glasgow and Belfast areas.
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measurement of successful device use (Flutiform® pMDI) versus (breath activated device (BAI)) | One day only for each device
  This study compares our Flutiform® pMDI (pressurised metered dose inhaler) containing placebo only and a breath activated device (BAI), containing placebo only. The percentage of subjects will be measured who have successful device use using an 8 point scale.

SECONDARY OUTCOMES:
The percentage of subjects able to generate an adequate inspiratory flow to trigger the BAI. | Each device will be used on one day only
The percentage of subjects with successful device use | Each device will be used for one day only
  This is defined as all critical steps being correctly performed - Steps 2, 4 - 6 for pMDI; Steps 2, 4 - 7 for BAI; on an 8 point scale
The percentage of subjects unable to be trained to use the device successfully within 15 minutes | Each device will be used on one day only
The percentage of subjects able to perform 7, 6, 5, 4, 3, 2, and 1 step successfully. | Each device will be used for one day only
  Measured on an 8 point scale

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - BioKinetic Europe Ltd, Belfast
  - Glasgow Clinical Research Facility, Glasgow

REFERENCES:
- [Derived] Bell D, Mansfield L, Lomax M. A Randomized, Crossover Trial Evaluating Patient Handling, Preference, and Ease of Use of the Fluticasone Propionate/Formoterol Breath-Triggered Inhaler. J Aerosol Med Pulm Drug Deliv. 2017 Dec;30(6):425-434. doi: 10.1089/jamp.2017.1385. Epub 2017 Jul 6. PMID 28683212